CLINICAL TRIAL: NCT06605794
Title: A Prospective, Multi-center Study to Evaluate the Safety and Efficacy of FreeFlow Percutaneous Atrial Septal Shunt in Patients With Idiopathic Pulmonary Arterial Hypertension
Brief Title: FreeFlow Percutaneous Atrial Septal Shunt for IPAH
Acronym: FREEFLOW
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-111R
Record Dates: First submitted 2024-08-20; First posted 2024-09-20 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Device-intervention Group (Experimental): FreeFlow percutaneous atrial septal shunt
  Interventions: Device: FreeFlow percutaneous atrial septal shunt

INTERVENTIONS:
Device: FreeFlow percutaneous atrial septal shunt — The trial devices included a percutaneous atrial septal shunt and an atrial septal shunt delivery system. The specifications of the atrial septal shunt device were -φ5, φ7, φ9, φ11, and the specifications of the atrial septal shunt delivery system-FFISS-B were 9F and 10F.

SUMMARY:
The goal of this clinical trial is to explore the safety and efficacy of the FreeFlow percutaneous atrial septal shunt for treatment of idiopathic pulmonary arterial hypertension. The main questions it aims to answer are:

* Is the FreeFlow percutaneous atrial septal shunt safe to use in patients with idiopathic pulmonary arterial hypertension?
* Does the FreeFlow percutaneous atrial septal shunt reduce all-cause mortality and readmission in patients with idiopathic pulmonary arterial hypertension, and how effective is it? Thirty subjects who met the inclusion and exclusion criteria were selected for selective implantation of FreeFlow percutaneous atrial septal shunts after balloon atrial septostomy.

Participants will:

* underwent balloon atrial septostomy and FreeFlow percutaneous atrial septal shunt implantation.
* will be followed up at 24 hours after shunt implantation or before discharge, 1 month, 3 months, 6 months and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* 18≤ age ≤70 years old, female or male;
* 10 mmHg≤ mean right atrial pressure (mRAP) ≤20 mmHg;
* The subjects had severe idiopathic pulmonary hypertension (mean pulmonary arterial pressure > 45 mmHg);
* WHO grade III or IV;
* NT-proBNP≥650 ng/L;
* The subjects were informed of the nature of the study and agreed to all the requirements for participating in the study. They signed the informed consent form and agreed to complete the follow-up and the examinations required for the follow-up.

Exclusion Criteria:

* Local or systemic sepsis or other acute infection;
* Severe coagulopathy;
* Allergy to nickel and/or titanium and/or nickel/titanium-based materials;
* Patients with contraindications to antiplatelet, coagulant or thrombotic therapy;
* Intolerance to contrast media;
* Have participated in other drug or device clinical trials during the same period;
* Glomerular filtration rate (GFR) < 50 mL/min;
* Patients with severe liver dysfunction (alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 3 times the upper limit of normal);
* The patient had malignant arrhythmia;
* The patient did not receive standardized drug therapy (triple sequential therapy) according to the Chinese guidelines for the diagnosis and treatment of pulmonary hypertension within 3 months;
* Women who are pregnant, planning to become pregnant (within 12 months) or breastfeeding;
* Severe restrictive or obstructive lung disease;
* Implanted atrial septal defect (ASD)/ patent foramen ovale (PFO) closure device;
* Left ventricular ejection fraction (LVEF) <50%;
* SpO2 < 90% without oxygen inhalation (pulse measurement);
* The anatomical structure of the heart is abnormal, and the shunt cannot be implanted on the atrial septum;
* Other circumstances in which the patient was deemed by the investigator to be ineligible for inclusion in the trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-09-11 (Actual); Primary Completion 2027-09-11 (Estimated); Study Completion 2027-09-11 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality at 6 months | 6 months
  All-cause mortality at 6 months
Rehospitalization rates associated with exacerbation of pulmonary arterial hypertension | 6 months
  Rehospitalization rates associated with exacerbation of pulmonary arterial hypertension within 6 months

SECONDARY OUTCOMES:
Effective shunt rate at the end point | 12 months
  Effective shunt was defined as the presence of intra-atrial shunt by echocardiography at 12 months after operation, and the diameter of the shunt was reduced by no more than 2mm compared with the diameter measured by echocardiography before discharge
Shunt Success rate | 12 months
  Successful shunt operation was defined as successful shunt implantation, normal morphology and position, and basically the expected shunt size under fluoroscopy.
The WHO functional class was changed 12 months after operation | 12 months
  The WHO functional class was changed 12 months after operation
Changes in NT-pro BNP at 12 months after surgery | 12 months
  Changes in NT-pro BNP at 12 months after surgery
The change of exercise capacity (6min walking test) was observed 12 months after operation | 12 months
  The change of exercise capacity (6min walking test) was observed 12 months after operation
The change of subjects' Kansas City Cardiomyopathy Quality of Life Questionnaire score at 12 months after surgery | 12 months
  The change of subjects' Kansas City Cardiomyopathy Quality of Life Questionnaire score at 12 months after surgery
Cumulative number of readmissions associated with exacerbation of pulmonary hypertension at 12 months after surgery | 12 months
  Cumulative number of readmissions associated with exacerbation of pulmonary hypertension at 12 months after surgery
Serious Adverse Event Rate (SAE) | through study completion, an average of 1 year
  Serious adverse event rate (SAE) refers to events occurring during the course of the clinical trial that lead to death or serious deterioration of health status, including fatal illness or injury, permanent defects in body structure or function, and the need for medical or surgical intervention to avoid permanent defects in body structure or function.
Device-related Adverse Event Rate (DSAE) | through study completion, an average of 1 year
  The device-related adverse event rate (DSAE) refers to the adverse medical events related to the use of the device that occurred during the course of the clinical trial.

CONTACTS AND LOCATIONS:
Overall Officials: Junbo GE, Prof., Principal Investigator — Fudan University
Locations (1):
- 180 Fenglin Road, Shanghai, Shanghai Municipality, China